CLINICAL TRIAL: NCT05602987
Title: The Effect of Enema on Postoperative Recovery and Complications in Anal Surgery: A Randomized Controlled Study
Brief Title: Comparison Study of the Effect of Enema in Anal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Tungcheng Chang, MD, PhD, Chief of Colorectal Surgery, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202209016
Record Dates: First submitted 2022-10-29; First posted 2022-11-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hemorrhoids; Fistula
MeSH Terms: conditions — Hemorrhoids; Fistula | interventions — Enema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group: enema (Experimental): receiving enema at the night before anal surgery
  Interventions: Procedure: enema
- Control Group: no enema (Active Comparator): no enema before anal surgery
  Interventions: Procedure: no enema

INTERVENTIONS:
Procedure: enema — receiving enema at the night before anal surgery
  Arms: Study Group: enema
Procedure: no enema — no enema before anal surgery
  Arms: Control Group: no enema

SUMMARY:
To evaluate whether receiving enema before anal surgery or not affects the postoperative recovery and complications.

DETAILED DESCRIPTION:
For patients undergoing anal surgery, some of them receive enema as doctors' preference before the surgery in consider to lower postoperative complications e.g. infection, while others do not. These choices are often determined by surgeons' personal preference according to their experiences due to lack of evidence from researches. Hemorrhoidectomy and fistulotomy are the most common two types of surgery in colon and rectal surgery division in Shuang Ho hospital, where top three quantities of hemorrhoidectomy in Taiwn have been performed.Therefore, we conducted a randomized controlled trial to evaluate the benefits of enema before anal surgery and possible waste of medical resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent hemorrhoidectomy, including circular stapled hemorrhoidopexy (PPH) and conventional hemorrhoidectomy
* Patients who underwent fistulotomy or fistulectomy

Exclusion Criteria:

* Emergency surgery
* Surgery other than circular stapled hemorrhoidopexy (PPH) and conventional hemorrhoidectomy, e.g., rubber band ligation, injection treatment, and cryosurgery
* Complicated fistulectomy, e.g., requiring surgical drainage and seton placement
* Other types of anal surgery, e.g., anal fissure and colorectal cancer
* Liver cirrhosis
* Coagulation dysfunction
* Bedridden
* Human immunodeficiency virus infection

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09-10 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pain score | On postoperative day 0 to day 7
  record max pain score(visual analog scale:0-10) each day
Consumption of analgesics | On postoperative day 0 to day 7
  daily consumption of oral analgesics from post-operative day 0 to day 7

SECONDARY OUTCOMES:
Incidence of surgical site infection | On postoperative day 0-30
  Surgical site infection was defined as hospital admission for infection management or need for surgical intervention to manage the wound.
Incidence of Urinary retention | On postoperative day 0 to day 7
  patients requiring foley catheterization during hospital stay
First defecation after surgery | On postoperative day 0 to day 7
  Time between first defecation and operation

CONTACTS AND LOCATIONS:
Overall Officials: Tung Cheng Chang, MD, PHD, Study Director — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang-Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets used in this study can be obtained from the investigator upon reasonable request.
Supporting Information: Study Protocol
Time Frame: data is available as the study is complete and for 12 month period
Access Criteria: will be shared upon request